CLINICAL TRIAL: NCT05814081
Title: How To Prevent Ventilator-Related Lung Damage in Intraoperative Mechanical Ventilation? Pcv or Vcv ?
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Furkan Tontu, Anesthesiologist, Anesthesiology and Reanimation Department, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 21-20-07
Record Dates: First submitted 2023-03-16; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Ventilator-Induced Lung Injury; Ventilator Lung; Mechanical Ventilation Complication; Postoperative Complications
Keywords: mechanical power; prone; supine; postoperative pulmonary complications
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Postoperative Complications; Deception | interventions — Patient Positioning; Ventilation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pressure Control Ventilation Supine Group: 20 patients were ventilated in the supine position with pressure control mode.
  Interventions: Procedure: Position/Ventilation
- Pressure Control Ventilation Prone Group: 20 patients were ventilated in the prone position with pressure control mode.
  Interventions: Procedure: Position/Ventilation
- Volume Control Ventilation Supine Group: 20 patients were ventilated in the supine position with volume control mode.
  Interventions: Procedure: Position/Ventilation
- Volume Control Ventilation Prone Group: 20 patients were ventilated in the prone position with volume control mode.
  Interventions: Procedure: Position/Ventilation

INTERVENTIONS:
Procedure: Position/Ventilation — Positioning and ventilation mode adjustments were made to the patients.

SUMMARY:
Introduction: Intraoperative Mechanical Ventilation practices can lead to ventilator-associated lung injury (VILI) and postoperative pulmonary complications in healthy lungs. Mechanical Power has been developed as a new concept in reducing the risk of postoperative pulmonary complications as it takes into account all respiratory mechanics that cause VILI formation. Volume control mode is at the forefront in the old anesthesia devices used in the operating room, and today, together with technology, there are anesthesia devices with many modes and features, as in intensive care units. This causes confusion in the use of mechanical ventilators. In this study, volume and pressure control ventilation modes were compared in terms of respiratory mechanics (including mechanical power) in patients operated in the supine and prone positions.

Aim of study: It has been compared the effects on postoperative pulmonary complications (PPH) in terms of VILI risk by calculating mechanical power from advanced respiratory mechanics of patients ventilated in pressure and volume control modes, which are frequently used in operating room applications.

Conclusion: There was no statistically significant difference between the groups in terms of demographic data, ariscat score, and ariscat risk group values. The supine and prone mechanical power (MPrs) values of the volume control group were statistically significantly lower than the pressure control group. P values were calculated as 0.012 and 0.001, respectively.

Results: Supine and prone MPrs values of the volume control group were calculated significantly lower than the pressure control group. Pressure-controlled intraoperative mechanical ventilation is considered to be disadvantageous in terms of the risk of VILI in the supine and prone position in terms of the current mechanical power concept.

DETAILED DESCRIPTION:
Although mechanical ventilation is a life-saving intervention, it can lead to ventilator-induced lung injury (VILI). VILI is the damage caused by positive pressure ventilation that starts with the use of mechanical ventilators. There are many factors that cause VILI such as tidal volume, drive pressure, flow, respiratory rate, and PEEP. Mechanical power, which collects these different variables in a single parameter, offers us new possibilities in predicting VILI at the bedside. The mechanical power being above a certain threshold causes damage ranging from pulmonary parenchymal rupture to severe inflammation and edema. Also, higher mechanical power values are associated with higher mortality. The protective ventilation strategy in intensive care units is also applied in operating rooms (OR) to minimize the risk of postoperative pulmonary complications due to VILI. While the volume control mode was at the forefront in the old anesthesia devices used in the OR, today there are anesthesia devices with many modes and features, as in intensive care units. This causes confusion in the use of mechanical ventilators in the perioperative period. Therefore, in this study, the investigators compared the perioperative mechanical power values in prone and supine positions, and postoperative pulmonary complications of two ventilation modes (volume control-pressure control ventilation). Thus, the investigators aimed to find out which ventilation mode would be advantageous in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - III risk group patients
* Patients between the ages of 18-70
* At least 2 hours of mechanical ventilation time

Exclusion Criteria:

* Patients with COPD or Asthma bronchial
* Patients with a functional capacity of less than 7 METS
* Pregnant and lactating female patients.
* Patients who have had thoracic surgery before
* Patients with BMI above 35
* Patients who had hemodynamic instability or desaturation (SpO2<92%) during the operation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cervical hernia, lumbar hernia and lumbar stabilization cases who were operated in the neurosurgery operating room of the anesthesia and reanimation clinic were examined.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Mechanical power | During surgery (2 hours to 4 hours)
  Mechanical power values calculated during surgery were compared.
Postoperative complications | Postoperative period (up to 10 days)
  Postoperative pulmonary complications were observed.

SECONDARY OUTCOMES:
Respiratory parameters other than mechanical power | During surgery (2 hours to 4 hours)
  PEEP(mmHg) value measured during surgery were compared.
Respiratory parameters other than mechanical power | During surgery (2 hours to 4 hours)
  Tidal volume(ml) value measured during surgery were compared.
Respiratory parameters other than mechanical power | During surgery (2 hours to 4 hours)
  Peak pressure(mmHg) value measured during surgery were compared.
Respiratory parameters other than mechanical power | During surgery (2 hours to 4 hours)
  Plato pressure(mmHg) value measured during surgery were compared.
Respiratory parameters other than mechanical power | During surgery (2 hours to 4 hours)
  Driving pressure(mmHg) value measured during surgery were compared.
Respiratory parameters other than mechanical power | During surgery (2 hours to 4 hours)
  Inspiratory time(second) value measured during surgery were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Furkan Tontu, Study Director — Basaksehir Cam & Sakura City Hospital
Locations (1):
- Basaksehir Cam Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet.

REFERENCES:
- [Result] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2013 Nov 28;369(22):2126-36. doi: 10.1056/NEJMra1208707. No abstract available. PMID 24283226
- [Result] Cressoni M, Gotti M, Chiurazzi C, Massari D, Algieri I, Amini M, Cammaroto A, Brioni M, Montaruli C, Nikolla K, Guanziroli M, Dondossola D, Gatti S, Valerio V, Vergani GL, Pugni P, Cadringher P, Gagliano N, Gattinoni L. Mechanical Power and Development of Ventilator-induced Lung Injury. Anesthesiology. 2016 May;124(5):1100-8. doi: 10.1097/ALN.0000000000001056. PMID 26872367
- [Result] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Result] Tonetti T, Vasques F, Rapetti F, Maiolo G, Collino F, Romitti F, Camporota L, Cressoni M, Cadringher P, Quintel M, Gattinoni L. Driving pressure and mechanical power: new targets for VILI prevention. Ann Transl Med. 2017 Jul;5(14):286. doi: 10.21037/atm.2017.07.08. PMID 28828361
- [Result] Giosa L, Busana M, Pasticci I, Bonifazi M, Macri MM, Romitti F, Vassalli F, Chiumello D, Quintel M, Marini JJ, Gattinoni L. Mechanical power at a glance: a simple surrogate for volume-controlled ventilation. Intensive Care Med Exp. 2019 Nov 27;7(1):61. doi: 10.1186/s40635-019-0276-8. PMID 31773328
- [Result] Asar S, Acicbe O, Cukurova Z, Hergunsel GO, Canan E, Cakar N. Bedside dynamic calculation of mechanical power: A validation study. J Crit Care. 2020 Apr;56:167-170. doi: 10.1016/j.jcrc.2019.12.027. Epub 2020 Jan 2. PMID 31931417